CLINICAL TRIAL: NCT04556422
Title: Standalone Sauna Versus Exercise Followed by Sauna on Cardiovascular Function in Non-naïve Sauna Users
Brief Title: Comparison of Acute Sauna With Exercise and Sauna
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: Finnish Foundation for Cardiovascular Research (Other); Business Finland (Other); Harvia Finland Oy (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Sauna
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Risk Factor; Blood Pressure; Arterial Stiffness
Keywords: Sauna bathing; Aerobic exercise; Thermal therapy; Passive heat
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sauna alone (Active Comparator): Sauna exposure for 30 minutes
  Interventions: Other: Sauna bathing
- Exercise and Sauna (Experimental): Cycling exercise for 15 minutes followed by sauna for 15 minutes
  Interventions: Other: Aerobic exercise; Other: Sauna bathing

INTERVENTIONS:
Other: Aerobic exercise — 15 minutes of aerobic exercise using stationary bicycle
  Arms: Exercise and Sauna
Other: Sauna bathing — Passive heat exposure

SUMMARY:
Sauna bathing has been associated with a lower risk for cardiovascular disease (CVD) outcomes, improved vascular endothelial and cardiac function, reduced oxidative stress and lower blood pressure. Earlier studies conducted by the investigators have showed positive alterations of arterial stiffness and hemodynamics through sauna bathing.

Some studies have sought to utilize sauna bathing as an intervention after exercise with promising and synergistic results, although the effects on populations with cardiovascular risk factors are less clear. Furthermore, studies investigating the use of both exercise and sauna bathing in combination has been somewhat limited. However, results from some studies speculate that adjunctive exercise and sauna interventions may be useful for aging and clinical patient population groups.

Given that heat therapy and sauna use is gaining more worldwide popularity, the investigators sought to compare the acute hemodynamic effects between sauna use alone and a short bout of exercise followed by sauna exposure. It was hypothesize that the combination of exercise and sauna will elicit greater changes than sauna alone. To achieve this, we standardized the protocol duration (30 minutes).

DETAILED DESCRIPTION:
In this crossover trial, all study participants underwent two interventions, each on a separate occasion (>72 hours apart). A standalone 30-minute sauna at 75°C (S), and 15-minutes of cycling on the stationary bike at 75% maximum heart rate, followed by 15-minutes of sauna exposure (ES). A cycling exercise test was conducted on a separate day prior to the experiment to ascertain individual maximal exercise heart rates, which was then used to calculate individual 75% maximum.

After the ﬁrst 15-minute period of S, the participants left the sauna room to have a quick shower (<30 seconds) before going back for the second 15-minute period. The same sauna bathing room (75°C) was used for all participants and the cycling exercise was conducted within 10 meters of the sauna room to minimize transit time during ES. Participants were instructed to abstain from eating 2h, caffeine 12h and alcohol 24h prior to the measurements. Food intake was not standardized. Fluid was consumed ad libitum. A medical physician was in attendance at all times and participants were allowed to leave the sauna or stop the experiment at any time if they felt uncomfortable.

Brachial blood pressures and pulse wave velocity (PWV) as a measure of arterial stiffness, were taken in their respective order at three different time points; before (PRE), immediately after (POST), and after a 30-minute recovery (POST30). Transit time from the cessation of the intervention to POST measurements were kept under 60 seconds. All measurements were performed by the same assessor to minimize ascertainment biases.

Participants were permitted to take a quick shower (<30 seconds) before POST measurements were taken. Water temperature or the shower was not controlled and participants could freely select their desired temperature. Thereafter, they were instructed to rest in a designated waiting lounge (mean temperature 21°C) in a seated position for a duration of 30-minutes before the last measurement (POST30) was taken.

ELIGIBILITY:
Inclusion Criteria:

* Free of a prior diagnosis of CVD, exhibits at least one of the following cardiovascular risk factors: a history of smoking, hyperlipidemia, hypertension, diabetes, obesity, or family history of coronary heart disease (CHD).

Exclusion Criteria:

* recent musculoskeletal injuries or surgery (less than 6 months ago), mental illnesses, under 30 years of age or over 75 at time of recruitment, health conditions that may contraindicate study parameters.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Brachial blood pressure | Single session (30 minutes)
  Systolic and diastolic blood pressure
Central blood pressure | Single session (30 minutes)
  Systolic and diastolic blood pressure measured using ECG and Pulsepen

SECONDARY OUTCOMES:
Arterial Stiffness | Single session (30 minutes)
  Pulsewave velocity (PWV)
Augmentation Index | Single session (30 minutes)
  Supplement to PWV

CONTACTS AND LOCATIONS:
Overall Officials: Jari A Laukkanen, PhD/MD, Principal Investigator — Central Finland Central Hospital
Locations (1):
- University of Jyväskylä, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee E, Laukkanen T, Kunutsor SK, Khan H, Willeit P, Zaccardi F, Laukkanen JA. Sauna exposure leads to improved arterial compliance: Findings from a non-randomised experimental study. Eur J Prev Cardiol. 2018 Jan;25(2):130-138. doi: 10.1177/2047487317737629. Epub 2017 Oct 19. PMID 29048215
- [Background] Laukkanen T, Kunutsor SK, Zaccardi F, Lee E, Willeit P, Khan H, Laukkanen JA. Acute effects of sauna bathing on cardiovascular function. J Hum Hypertens. 2018 Feb;32(2):129-138. doi: 10.1038/s41371-017-0008-z. Epub 2017 Dec 21. PMID 29269746
- [Background] Lee E, Willeit P, Laukkanen T, Kunutsor SK, Zaccardi F, Khan H, Laukkanen JA. Acute effects of exercise and sauna as a single intervention on arterial compliance. Eur J Prev Cardiol. 2020 Jul;27(10):1104-1107. doi: 10.1177/2047487319855454. Epub 2019 Jun 8. No abstract available. PMID 31177835